CLINICAL TRIAL: NCT01901211
Title: CP Fit 'n' Fun Project: Physical and Social Benefits of Multi-Player Interactive Computer Play Games in Youth With Cerebral Palsy
Brief Title: Physical and Social Benefits of Multi-Player Interactive Computer Play Games in Youth With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: Queen's University (Other); Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 13-423
Record Dates: First submitted 2013-07-11; First posted 2013-07-17 (Estimated); Results first posted 2017-03-17 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2016-01

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Interactive computer play; Multi-player gaming; Exercise
MeSH Terms: conditions — Cerebral Palsy; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exergaming (Experimental): In this arm, the participants will participate in the exergaming intervention.
  Interventions: Other: Exergaming Intervention
- Comparison Arm (No Intervention): In this arm of the study, participants will engage in their typical physical activity routines for the ten week duration. Participants will receive a call from the RA each week. The RA will ask the child to report on all the physical and social activities that they engaged in for that week.

INTERVENTIONS:
Other: Exergaming Intervention — The exergaming system will be installed into the participants' homes. Players will pedal the exergame bike in order to move their game avatar. Headsets allow players to communicate with each other in real-time. Participants will play the games 3 to 5 times per week, during scheduled game times. Players will wear a heart rate (HR) monitor and will achieve game benefits for reaching their target HR. They will be asked to exercise in a target HR zone of 40-65%HR reserve. Each week, participants will receive a call from a research assistant (RA), who will provide feedback on their exercise progress and a HR goal for each week. The RA will also record physical and social activities engaged in and any difficulties like leg pain or technical issues.
  Arms: Exergaming

SUMMARY:
As children with cerebral palsy (CP) become teenagers, they experience a decrease in their physical function and mobility. Decreased mobility leads to increased social isolation for the teens and impacts negatively on their quality of life. This loss of function is multifactorial, but poor physical fitness and muscle weakness secondary to disuse are significant contributors. Exercise video games are a novel approach to engage youth in physical exercise and social interaction with their peers. The objective of this study is to evaluate the impact of an exercise video gaming intervention to improve physical fitness and social wellbeing. Our over-arching research questions are whether "exergames" can provide health benefits (improved physical fitness) and improved social wellbeing in youth with CP.

DETAILED DESCRIPTION:
The primary objectives of this study are to evaluate the impact of exergaming on cardiovascular fitness and social wellbeing related to friends/peers in youths with CP. The secondary objectives of the study will be to evaluate the impact of the exergaming intervention on additional components of physical fitness including anaerobic fitness, and muscle strength. In addition, the effect of the exergaming intervention on overall health-related quality of life (HRQL), self-esteem and motor participation will also be measured. Finally, the effectiveness of a technique for balancing performance in multiplayer exergames will be evaluated. The objectives will be investigated using a randomized crossover study design.Outcomes will be measured a total of four times: at study entry and after the first ten-week period (either comparison or intervention), at the end of a six-week washout period, then again after second period (either intervention or comparison). Outcomes will be assessed by physiotherapists and research staff members who will be blinded to the condition of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CP and GMFCS level III
* Between 9 and 18 years of age inclusive
* Ability to operate a handheld videogame controller
* High-speed internet in the home
* Able to commit for the entire study duration

Exclusion Criteria:

* Orthopedic surgery in the preceding six months
* Exercise-induced asthma
* Any underlying heart condition
* Seizure disorder
* Visual, auditory or cognitive disabilities that will interfere with game play

Ages: 9 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2014-04-05 (Actual); Study Completion 2014-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darcy Fehlings, MD, MSc, FRCPC, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital; T.C. Nicholas Graham, PhD, Principal Investigator — Queen's University
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Exergaming First, Then Comparison: In this arm, the participants will participate in the exergaming intervention during the first ten-week period then after 6-week washout, will participate in the comparison during the second ten-week period.
  Exergaming Intervention: The exergaming system will be installed into the participants' homes. Players will pedal the exergame bike in order to move their game avatar. Headsets allow players to communicate with each other in real-time. Participants will play the games 3 to 5 times per week, during scheduled game times. Players will wear a heart rate (HR) monitor and will achieve game benefits for reaching their target HR. They will be asked to exercise in a target HR zone of 40-65%HR reserve. Each week, participants will receive a call from a research assistant (RA), who will provide feedback on their exercise progress and a HR goal for each week. The RA will also record physical and social activities engaged in and any difficulties like leg pain or technical issues.
- Comparison First, Then Exergaming: In this arm of the study, participants will participate in comparison activities during the first ten-week period then after 6-week washout, will participate in the Exergaming activities during the second ten-week period.
  participants will engage in their typical physical activity routines for the ten week duration. Participants will receive a call from the RA each week. The RA will ask the child to report on all the physical and social activities that they engaged in for that week.
Period: First Ten-week Period
Arm/Group | Exergaming First, Then Comparison | Comparison First, Then Exergaming
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Washout (6 Weeks)
Arm/Group | Exergaming First, Then Comparison | Comparison First, Then Exergaming
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Second Ten-week Period
Arm/Group | Exergaming First, Then Comparison | Comparison First, Then Exergaming
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Exergaming First, Then Comparison: In this arm, the participants will participate in the exergaming intervention during the first ten-week then after 6-week washout, will participate in the comparison activities during the second ten-week period.
  Exergaming Intervention: The exergaming system will be installed into the participants' homes. Players will pedal the exergame bike in order to move their game avatar. Headsets allow players to communicate with each other in real-time. Participants will play the games 3 to 5 times per week, during scheduled game times. Players will wear a heart rate (HR) monitor and will achieve game benefits for reaching their target HR. They will be asked to exercise in a target HR zone of 40-65%HR reserve. Each week, participants will receive a call from a research assistant (RA), who will provide feedback on their exercise progress and a HR goal for each week. The RA will also record physical and social activities engaged in and any difficulties like leg pain or technical issues.
- Comparison First, Then Exergaming: In this arm of the study, participants will complete comparison activities during the first ten-week then after 6-week washout, will participate in the exergaming intervention during the second ten-week period.
  Participants will engage in their typical physical activity routines for the ten week duration. Participants will receive a call from the RA each week. The RA will ask the child to report on all the physical and social activities that they engaged in for that week.
- Total: Total of all reporting groups
Arm/Group | Exergaming First, Then Comparison | Comparison First, Then Exergaming | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 4 | 10
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.5 (1.3) | 16.0 (2.4) | 15.2 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 4 | 4 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in the 7.5 Meter Shuttle Run Test for Gross Motor Function Classification Scale (GMFCS) Level III (SRT-III)
Description: The 7.5m Shuttle Run test (SRT-III) is a maximal, running-based, field test that can assess cardiovascular fitness in children with CP GMFCS level III. In the tests, markers are placed 7.5m apart in a square formation. Participants walk from marker to marker according to progressively faster auditory cues from a music device. The assessment is scored by the total number of shuttle run levels that the participant completes to the nearest half shuttle. A higher score is better.
Time Frame: Baseline (1-week pre-study arm 1), 11-weeks (post study arm 1), 17-weeks (post washout period), 28-weeks (post study arm 2)
Population: One participant was unable to complete post-assessment after Exergaming Arm. Therefore, 11 participants did complete the protocol, as indicated in the participant flow section, however change scores for outcome measures were not calculated for one participant during the Exergaming Arm. This participant was part of the Comparison First group.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Exergaming: In this arm, the participants will participate in the exergaming intervention in either the first or the last part of the study.
  Exergaming Intervention: The exergaming system will be installed into the participants' homes. Players will pedal the exergame bike in order to move their game avatar. Headsets allow players to communicate with each other in real-time. Participants will play the games 3 to 5 times per week, during scheduled game times. Players will wear a heart rate (HR) monitor and will achieve game benefits for reaching their target HR. They will be asked to exercise in a target HR zone of 40-65%HR reserve. Each week, participants will receive a call from a research assistant (RA), who will provide feedback on their exercise progress and a HR goal for each week. The RA will also record physical and social activities engaged in and any difficulties like leg pain or technical issues.
- Comparison Arm: In this arm of the study, participants will engage in their typical physical activity routines for the ten week duration in either the first or the last part of the study.
  Participants will receive a call from the RA each week. The RA will ask the child to report on all the physical and social activities that they engaged in for that week.
Arm/Group | Exergaming | Comparison Arm
Number analyzed (Participants) | 10 | 11
units on a scale
  SRT at baseline | 8.3 (7.2) | 8.6 (6.4)
  SRT change from baseline | 1.1 (1.7) | 0.7 (2.6)

2. Primary Outcome: Change in the Social Wellbeing Domain of the KINDL-R Quality of Life Questionnaire
Description: Wellbeing Related to Friends/Peers domain of the KINDL-R is a four-item subscale focusing on time spent with friends, being perceived as a success with friends, getting along with friends and whether or not they felt different from peers over the past week.
  The subscale has 4 items scored on a five-point Likert scale that can be scored in isolation and is converted to percent of total subscale score. Full range of possible scores 0-20. Score is converted to percent of total subscale score (0-100%). Higher scores indicate greater social wellbeing.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of total subscale score
Arm/Group | Exergaming | Comparison Arm
Number analyzed (Participants) | 10 | 11
percentage of total subscale score
  Social Wellbeing Domain of the KINDL-R at baseline | 63.1 (26) | 79.4 (23.1)
  Social Wellbeing Domain of the KINDL-R change | 14.4 (25.3) | -5.6 (24.1)

3. Secondary Outcome: Handheld Dynamometry Measures of Knee Flexors and Knee Extensors
Description: Handheld dynamometry will be used to measure muscle strength for the quadriceps muscles and the hamstrings at 90˚ of knee flexion in both legs.
  The individual sits with legs at 90˚ of knee flexion and resistance will be given anteriorly (knee extensors) and posteriorly (knee flexors) two inches proximal to the lateral malleoli.
  Higher score indicates greater strength.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Exergaming | Comparison Arm
Number analyzed (Participants) | 10 | 11
pounds
  Quad-Left at baseline | 12.1 (6.1) | 11.5 (4.6)
  Quad-Left change from baseline | -0.1 (5.4) | 0.1 (3.5)
  Quad-Right at baseline | 11.5 (4.4) | 11.5 (4.4)
  Quad-Change change from baseline | -0.8 (4.4) | 0.1 (3.2)
  Hamstring-Left at baseline | 4.9 (4.4) | 5.2 (4.0)
  Hamstring-Left change from baseline | 0.5 (2) | 1.3 (1.5)
  Hamstring-Right at baseline | 5.5 (3.8) | 5.3 (3.8)
  Hamstring-Right change from baseline | 0.2 (2.7) | 0.8 (2.0)

4. Secondary Outcome: The 30-second Wingate Cycle Test
Description: The 30-second Wingate Cycle Test is a measure of anaerobic power, a key component of physical fitness. The cycle test is performed when a participant uses a cycle ergometer and pedals as hard as they can for 30-seconds against a constant braking force.
  The measure is relative peak power (watts/kg) normalized to body weight. Higher scores indicate greater anaerobic power.
Time Frame: as for outcome 1
Population: This test was unsuitable for over half the participants, who were unable to complete one or more of the 30-second Wingate tests. Malfunctioning equipment also made collecting full data sets impossible.
Measure: Mean (Standard Deviation); unit: Watts/Kg
Arm/Group | Exergaming | Comparison Arm
Number analyzed (Participants) | 5 | 5
Watts/Kg
  Relative peak power baseline | 1.92 (1.54) | 2.49 (1.41)
  Relative peak power change | 0.26 (1.0) | -0.01 (1.43)

5. Secondary Outcome: Anthropometric Measurements
Description: Anthropometric measurements of waist circumference, triceps and subscapular skinfold thickness, will be used to assess body composition as indicators of physical fitness.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Exergaming | Comparison Arm
Number analyzed (Participants) | 10 | 11
cm
  Waist circumference at baseline | 83.2 (14.4) | 80.1 (14.4)
  waist circumference change from baseline | -1.2 (1.6) | 2.5 (2.5)
  Tricep skinfold thickness at baseline | 2.67 (10.52) | 15.60 (8.13)
  Tricep skinfold thickness change from baseline | -0.93 (4.70) | 0.85 (5.04)
  Subscap skinfold thickness at baseline | 13.67 (5.77) | 11.87 (14.40)
  Subscap skinfold thickness change from baseline | 2.08 (2.08) | 6.90 (12.97)

6. Secondary Outcome: Total Score of the KINDL-R Questionnaire
Description: The total score of the 24-item KINDL-R questionnaire will measure the participants' health-related quality of life.
  Scores are on a five-point Likert scale that can be scored in isolation and is converted to percent of total score. Total score is the summed score divided by the total possible score. Full range of possible scores 0-120. Score is converted to percent of total subscale score (0-100%). Higher scores indicate greater health related quality of life.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of total score on a scale
Arm/Group | Exergaming | Comparison Arm
Number analyzed (Participants) | 10 | 11
percentage of total score on a scale
  Total Score of the KINDL-R at baseline | 68.3 (8.1) | 73.3 (14.2)
  Total Score of the KINDL-R change from baseline | 2 (12.8) | -7.4 (17.1)

7. Secondary Outcome: The Self-Worth Domain of the KINDL-R Questionnaire
Description: The 4-item Self-worth Domain of the KINDL-R will be used as an indicator of self-esteem.
  The subscale has 4 items scored on a five-point Likert scale that can be scored in isolation and is converted to percent of total subscale score. Full range of possible scores 0-20. Score is converted to percent of total subscale score (0-100%). Higher scores indicate greater self-worth.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of total subscale score
Arm/Group | Exergaming | Comparison Arm
Number analyzed (Participants) | 10 | 11
percentage of total subscale score
  KINDL-R at baseline | 69.4 (19.5) | 77.5 (19.4)
  KINDL-R change from baseline | 3.1 (21.5) | -10.6 (26.5)

8. Secondary Outcome: Gaming Data
Description: Gaming data will be collected as measures of effectiveness of the games' balancing techniques, engagement and adherence. The games will be instrumented to automatically collect usage data including: amount of time playing; amount of time within HR zones while playing.
  Higher numbers indicate more activity and more time above 40% hear rate reserve (HRR) while playing.
Time Frame: 10-weeks of the exergaming intervention
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Exergaming
Number analyzed (Participants) | 11
minutes
  Minutes above 40% Heart Rate Reserve per day | 14.7 (8.8)
  Minutes of activity from exergame per day | 35.4 (10.9)

9. Secondary Outcome: StepWatch Activity Monitors
Description: StepWatch Activity Monitors will be used to measure activity levels and motor participation. The StepWatch is a two-plane accelerometer that is worn around the ankle in a knit cuff. The StepWatch measures ambulatory activity (i.e. total daily step count) and acts as an indicator of motor participation in the community.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Steps/day
Arm/Group | Exergaming | Comparison Arm
Number analyzed (Participants) | 10 | 10
Steps/day
  StepWatch Activity at baseline | 77.5 (69.5) | 86.1 (96.4)
  StepWatch Activity change from baseline | 21.3 (55.2) | -21.0 (63.3)

10. Secondary Outcome: Anthropometric Measurements (Weight)
Description: Anthropometric measurements of waist circumference, triceps and subscapular skinfold thickness, and weight will be used to assess body composition as indicators of physical fitness.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Exergaming | Comparison Arm
Number analyzed (Participants) | 10 | 11
Kg
  Weight at baseline | 52.2 (23.4) | 47.2 (14.4)
  Weight change from baseline | -2.5 (17.5) | 0.8 (5.7)

ADVERSE EVENTS:
Groups:
- Exergaming: In this arm, the participants will participate in the exergaming intervention during the first ten-week period then after 6-week washout, will participate in the comparison during the second ten-week period.
  Exergaming Intervention: The exergaming system will be installed into the participants' homes. Players will pedal the exergame bike in order to move their game avatar. Headsets allow players to communicate with each other in real-time. Participants will play the games 3 to 5 times per week, during scheduled game times. Players will wear a heart rate (HR) monitor and will achieve game benefits for reaching their target HR. They will be asked to exercise in a target HR zone of 40-65%HR reserve. Each week, participants will receive a call from a research assistant (RA), who will provide feedback on their exercise progress and a HR goal for each week. The RA will also record physical and social activities engaged in and any difficulties like leg pain or technical issues.
- Comparison Arm: In this arm of the study, participants will participate in comparison activities during the first ten-week period then after 6-week washout, will participate in the Exergaming activities during the second ten-week period.
  participants will engage in their typical physical activity routines for the ten week duration. Participants will receive a call from the RA each week. The RA will ask the child to report on all the physical and social activities that they engaged in for that week.
Arm/Group | Exergaming | Comparison Arm
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 1/11 | 2/11
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exergaming (N=11) | Comparison Arm (N=11)
lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — lower back pain due to seat configuration (narrow or relation between seat and pummel)
Muscle soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — gluteus maximus muscle soreness
muscle soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (8) — quadriceps muscle tightness
Discomfort (Product Issues) | 0 (0) | 1 (1) — participant informed RA of headsets being uncomfortable and causing pain in ear

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No